CLINICAL TRIAL: NCT04044560
Title: Blinatumomab for Minimal Residual Disease (MRD) in Pre-B Cell Acute Lymphoblastic Leukemia Patients Following Hematopoietic Cell Transplantation: A Canadian, Multicentre Trial
Brief Title: Blinatumomab for MRD in Pre-B ALL Patients Following Stem Cell Transplant
Acronym: OZM-097
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrolment, loss of funding
Sponsor: University of British Columbia (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, David Sanford, Clinical Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H19-00893; CTTC 1902 (Other: Sponsor Protocol No.)
Record Dates: First submitted 2019-07-31; First posted 2019-08-05 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: B-cell Adult Acute Lymphoblastic Leukemia; Stem Cell Leukemia; Minimal Residual Disease
Keywords: acute lymphoblastic leukemia, blinatumomab, minimal residual disease, stem cell transplant
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Neoplasm, Residual; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Intervention Model Description: Participants will be monitored for MRD post transplant during the testing phase of the trial. If they have detectable MRD, they will be enrolled into the blinatumomab treatment phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Blinatumomab Treatment (Experimental): Eligible patients with detectable MRD will taper immunosuppressive medications, if applicable, and undergo treatment with blinatumomab. The duration of each cycle of blinatumomab treatment is 6 weeks. Adult and pediatric patients will be treated for 4 weeks followed by a 2-week treatment free period. Patients may receive up to 4 cycles total of blinatumomab therapy.
  Interventions: Biological: blinatumomab

INTERVENTIONS:
Biological: blinatumomab — Continuous intravenous infusion

SUMMARY:
This is a single arm, open label, multi-centre phase II study using blinatumomab for treatment of detectable minimal residual disease (MRD) in the first year following allogeneic hematopoietic stem cell transplant (HSCT) for patients with B cell acute lymphoblastic leukemia (B-ALL). The study has 2 phases: 1. MRD testing phase and 2. blinatumomab treatment phase. Participants with B-ALL planning for HSCT meeting other eligibility criteria will be enrolled onto the MRD testing phase, which will involve centralized MRD testing of bone marrow aspirate samples on day +56, +100, +180, +270 following HSCT. Participants with detectable MRD ≥10^-4 leukemic cells/total nucleated cells will enroll onto the treatment phase. Blinatumomab treatment will be started following detection of MRD after 7 to 42 days from enrollment onto the treatment phase to allow for initiation of taper of immunosuppressive medications.

ELIGIBILITY:
Testing Phase of Trial:

Inclusion Criteria:

* Pre-B-ALL in complete remission (CR), <5% blasts on most recent bone marrow aspirate determined by morphologic assessment, with an intention to proceed to allogeneic HSCT. Eligible participants can be in 1st CR or greater. Presence of detectable MRD by flow cytometry or other techniques in patients that are in morphologic remission prior to transplant is permitted.
* Detectable MRD measured by flow cytometry or other molecular techniques is acceptable for enrollment in patients with <5% blasts.
* Patients with either Philadelphia chromosome positive or negative B-ALL are eligible
* Documented expression of CD19 on the lymphoblast population as measured by flow-cytometry if patient has received prior CD19-directed therapy.
* Eligibility for HSCT along with conditioning regimen and donor selection will be determined according to the treating centre's policy.
* Patients must be age ≥1 years and have a baseline performance status of ECOG ≤ 2 (adult) or Lansky ≥ 50% (pediatric).
* Patient with chronic hepatitis B (Hep B surface antigen or Hep B Core antibody reactive) are eligible if they are receiving treatment to prevent reactivation (e.g. lamivudine, tenofovir) and have undetectable serum Hepatitis B DNA
* Patients (or legally acceptable designate) must provide written consent.
* Female patients of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study from the time of informed consent signature date until 3 months after completion of study treatment. Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

Exclusion Criteria:

* Inability to comply with study procedures.
* Active central nervous system (CNS) involvement or other extramedullary disease at the time of enrollment.
* Uncontrolled infection until resolved.
* Burkitt lymphoma/leukemia or mixed phenotype leukemia.
* Chronic infection with Hepatitis C. Previously treated Hepatitis C with undetectable Hepatitis C RNA for six months or longer is acceptable.
* HIV 1/2 Infection.

Treatment Phase of Trial:

Inclusion Criteria:

* Detectable MRD ≥ 10^-4 leukemic cells/TNC on a bone marrow aspirate done on day +56, +100, +180 or day +270.
* Morphologic remission on bone marrow from same date (on day +56, +100, +180 or day +270)
* Patients must be age ≥1 years and have a baseline performance status of ECOG ≤ 2 (adult) or Lansky ≥ 50% (pediatric) documented within 7 days of enrollment.
* Patients with either Philadelphia chromosome positive or negative B-ALL are eligible
* Documented expression of CD19 on the lymphoblast population as measured by flow-cytometry if patient has received prior CD19-directed therapy.
* Patient with chronic hepatitis B (Hep B surface antigen or Hep B Core antibody reactive) are eligible if they are receiving treatment to prevent reactivation (e.g. lamivudine, tenofovir) and have undetectable serum Hepatitis B DNA
* Adequate organ, liver and renal function including: Total bilirubin ≤ 1.5 x upper limit of normal (ULN), eGFR >30 mL/min/1.73 m, Alkaline phosphatase ≤ 2.5 x ULN, Serum lipase ≤ 1.5 x ULN
* Patients (or legally acceptable designate) must provide written consent.

Exclusion Criteria:

* Active acute GVHD (grade II-IV) or active moderate-severe chronic GVHD (NIH Grade) at the time of MRD detection are ineligible treatment phase until GVHD resolves or quiescent as determined by the treating physician.
* Uncontrolled infection until resolved.
* Chronic infection with Hepatitis C. Previously treated Hepatitis C with undetectable Hepatitis C RNA for six months or longer is acceptable.
* HIV 1/2 Infection.
* Extramedullary or CNS disease or the time of MRD detection.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
MRD Response | Following 1st cycle of blinatumomab (each cycle is 28 days)
  To determine the proportion of patients with MRD response, defined as negative MRD as measured by flow cytometry, after 1 cycle of blinatumomab.

SECONDARY OUTCOMES:
Safety and Tolerability | During Blinatumomab treatment, an average of 24 weeks
  Safety of delivering blinatumomab will be monitored early during the post-transplant course. Safety will be evaluated by the onset of treatment emergent adverse events (TEAEs) and by documentation of the incidence and severity of acute and chronic graft versus host disease (GvHD).
Survival | Up to 5 years
  Clinically relevant survival outcomes for patients enrolled onto the study including: 2-year and 5-year overall survival (OS) and event free-survival (EFS) and median OS.
Incidence of MRD Post HSCT | Up to day +270 following stem cell transplant
  To determine the proportion of patients developing detectable MRD following HSCT for B-ALL as measured by flow cytometry.
Patient Recruitment (Number of Patients Recruited) | Through Study Completion, an average of 2 years
  Feasibility
Turnaround time of centralized MRD testing (days) | Through Study Completion, an average of 2 years
  Feasibility
Time to delivery of blinatumomab following MRD detection | Through Study Completion, an average of 2 years
  Feasibility

CONTACTS AND LOCATIONS:
Overall Officials: David Sanford, MD, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - Vancouver General Hospital - Leukemia/Bone Marrow Transplant Program, Vancouver, British Columbia
  - BC Children's Hospital, Vancouver, British Columbia
  - QEII - Health Sciences Centre, Halifax, Nova Scotia